CLINICAL TRIAL: NCT03223077
Title: Mucosal and Microbiota Changes During Acute Campylobacteriosis
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 14-006180
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Post infectious
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Coded blood, stool (or other tissue) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Campylobacter: We will enroll 150 patients with acute Campylobacter infection. Our microbiology laboratory will inform us of a culture or PCR positive case of Campylobacter infection as soon as that test result is available.

SUMMARY:
Gastrointestinal (GI) infection with Campylobacter causes inflammation in the bowel and can change bacteria in the gut. Certain individuals with Campylobacter infection are also known to develop chronic bowel problems such as Irritable Bowel Syndrome (IBS). The researchers are doing this study to understand if changes in gut bacteria and gut mucosal lining during an acute infection can help identify individuals who might be at risk for developing problems in the future.

DETAILED DESCRIPTION:
Gastrointestinal (GI) infections involving a variety of bacterial, viral, and parasitic pathogens predispose patients to post-infectious irritable bowel syndrome (PI-IBS) and other functional GI disorders1. Campylobacter is one of the top five organisms responsible for food-borne illnesses causing approximately 0.8 million cases annually2. Isolated C. jejuni infection has been associated with a PI-IBS risk of 9% to 13%3. Epidemiological studies have identified female gender, age <60 years, smoking, enteritis severity, and pre-enteritis psychological stress as risk-factors for development of PI-IBS4. In a single study, variants in host genes TLR9, IL6, and CDH1 were identified as independent risk factors for development of PI-IBS after controlling for previously identified clinical risk factors5. In another study, host cytokines were looked at in relation to development of reactive arthritis and IBS following Campylobacter enteritis. The risk of acquiring clinical gastroenteritis with Campylobacter jejuni/coli was related to the INFG (+ 874A>T) of intron 1. Polymorphisms in IL-18 and INFG were linked to the risk of post-infectious reactive arthritis, but not to PI-IBS6. However, this study was limited by assessment of only serum cytokine profile and not mucosal. A recent study has shown that fecal microbiota of patients with PI-IBS differs from that of healthy controls and resembles that of patients with IBS with diarrhea (IBS-D)7. The microbiota is altered during acute enteritis, but it is unclear if there are any signatures in acute microbiota alterations that can help predict development of PI-IBS following Campylobacter enteritis. Our overall goal with this study is to identify non-invasive and invasive host factors that can help predict the development of PI-IBS following Campylobacter enteritis.

ELIGIBILITY:
Inclusion Criteria:

* No abdominal surgery (except appendectomy and cholecystectomy)
* Stool culture or Polymerase chain reaction (PCR) positive enteritis with Campylobacter

Exclusion Criteria:

* History of IBS, Irritable Bowel Disease (IBD) (Crohn's disease or ulcerative colitis), microscopic colitis or celiac disease.
* History of gastroenteritis in six months prior to Campylobacter enteritis
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute Campylobacter infection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-10-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Development of IBS is the endpoint. | 6 months
  Number of Subjects Who Develop Irritable Bowel Syndrome After Campylobacter Infection

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials